CLINICAL TRIAL: NCT01474759
Title: Portion Size Strategies for Management of Body Weight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Barbara J. Rolls, Principal Investigator, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PortionSize101; R01DK059853 (NIH)
Record Dates: First submitted 2011-11-15; First posted 2011-11-18 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Nutrition Assessment; Exercise; Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Portion size instruction (Experimental): Advice on diet, physical activity, and behavior change. Instruction in food portion size.
  Interventions: Behavioral: Advice on diet, physical activity, and behavior change; Behavioral: Instruction in food portion size
- Pre-portioned foods (Experimental): Advice on diet, physical activity, and behavior change. Provision of pre-portioned foods.
  Interventions: Behavioral: Advice on diet, physical activity, and behavior change; Other: Provision of pre-portioned foods
- Comparison (Active Comparator): Advice on diet, physical activity, and behavior change. Advice on healthy eating for weight loss.
  Interventions: Behavioral: Advice on diet, physical activity, and behavior change; Behavioral: Advice on healthy eating for weight loss

INTERVENTIONS:
Behavioral: Advice on diet, physical activity, and behavior change — Individuals will participate in individual sessions with Registered Dietitians providing basic instruction in principles of weight loss. The program will instruct individuals on the principles of healthy eating and nutrition during calorie restriction. These materials include one module with general information on the importance of limiting portion sizes. The program will also include instruction on physical activity and behavioral strategies for weight loss.
Behavioral: Instruction in food portion size — Individuals assigned to this program will participate in individual instructional sessions with specialized materials and tools that address food selection and choosing appropriate portion sizes of various foods.
  Arms: Portion size instruction
Other: Provision of pre-portioned foods — Individuals assigned to this program will be provided with commercially available pre-portioned foods and will be taught effective ways to incorporate them into their daily diet.
  Arms: Pre-portioned foods
Behavioral: Advice on healthy eating for weight loss — Individuals assigned to this program will participate in individual instructional sessions that address principles of healthy eating while on a calorie-restricted diet.
  Arms: Comparison

SUMMARY:
The primary aim of this research is to determine the efficacy of two portion-control strategies to achieve sustainable dietary and behavior changes and to promote weight loss and maintenance. A randomized controlled trial will test two approaches to managing portion sizes: one that gives individuals skills and tools to help them make appropriate portion choices, and another that focuses on consumption of pre-portioned foods in order to limit exposure to large portions in the personal food environment. A third group will receive a basic nutritional program to promote weight loss.

The second aim of the research is to determine the effects of the programs on knowledge and consumption of appropriate portions, as assessed by innovative assessment methods and multiple-pass dietary recalls. The third aim is to conduct exploratory analyses of individual factors that may influence the response to the portion-control interventions, such as psychosocial indicators, blood biomarkers, and measures of adherence to the interventions. The expected outcome of the project is that it will lead to the development of specific, evidence-based strategies to help control portion sizes in order to manage weight.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index of 28 to 45 kg/m squared
* Able to safely engage in physical activity (walking)
* Able to attend regular instructional sessions at University Park, Pennsylvania

Exclusion Criteria:

* have a medical condition diagnosed by a physician that precludes participation
* report symptoms indicative of depression or disordered eating
* report serious food allergies or intolerance
* current or planned participation in a weight-loss program
* pregnant or lactating or planning to become pregnant in the next 18 months

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2012-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in body weight | Months 0 to 12
  Body weight will be measured at multiple time points during the 12-month trial; the main outcome will be the weight trajectory across this time

SECONDARY OUTCOMES:
Change in portion size selection, perception, and knowledge | Months 0, 3, 6, & 12
  Computerized assessment of various foods (for self-selected portion sizes, estimation of calorie content, and satiety value) and general knowledge about portion size
Change in portion size consumption | Months 0, 3, 6, & 12
  Portion sizes consumed in various food categories as assessed by diet recalls and diet records
Change in blood biomarkers | Months 0, 3, 6, & 12
  Fasting lipids, glucose, insulin, and calculated insulin resistance
Change in waist circumference | Months 0, 3, 6, & 12
Change in blood pressure | Months 0, 3, 6, & 12
Change in dietary intakes | Months 0, 3, 6, 9, & 12
  Energy intake, nutrient intakes, dietary energy density, food group intakes, and diet quality from three days of 24-hour diet recalls
Change in step counts | Months 0, 3, 6, 9, & 12
  Daily step counts from pedometers
Change in attitudes and behaviors related to food and eating | Months 0, 1, 3, 6, & 12
  Self-reported eating attitudes and behaviors on multiple questionnaires
Change in psychosocial characteristics | Months 0, 3, 6, & 12
  Questionnaires measuring psychosocial characteristics including impulsivity, variety-seeking, and self-efficacy
Intervention adherence | Month 12
  Number of sessions attended, number of diet and activity records completed, and frequency of using intervention strategies during the entire trial

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J. Rolls, PhD, Principal Investigator — Penn State University
Locations (1):
- Penn State University Laboratory for the Study of Human Ingestive Behavior, University Park, Pennsylvania, United States

REFERENCES:
- [Derived] Roe LS, Rolls BJ. Which strategies to manage problem foods were related to weight loss in a randomized clinical trial? Appetite. 2020 Aug 1;151:104687. doi: 10.1016/j.appet.2020.104687. Epub 2020 Mar 29. PMID 32234531
- [Derived] James BL, Loken E, Roe LS, Rolls BJ. The Weight-Related Eating Questionnaire offers a concise alternative to the Three-Factor Eating Questionnaire for measuring eating behaviors related to weight loss. Appetite. 2017 Sep 1;116:108-114. doi: 10.1016/j.appet.2017.04.023. Epub 2017 Apr 22. PMID 28442337